CLINICAL TRIAL: NCT00269321
Title: Randomized Clinical Trial of Chiropractic Manual Therapy Plus Home Exercise, Supervised Exercise Plus Home Exercise and Home Exercise Alone For Individuals 65 and Over With Chronic Mechanical Low Back Pain
Brief Title: Chiropractic and Exercise for Seniors With Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Berman Center for Outcomes and Clinical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R18HP01424
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Low Back Pain
Keywords: Randomized; Clinical Trial; Low Back Pain; Chiropractic; Manual Therapies; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Procedure: Chiropractic Manual treatment + home exercise (procedure+behavior)
- 2 (Experimental)
  Interventions: Procedure: Supervised rehabilitative exercise+home exercise
- 3 (Active Comparator)
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Procedure: Chiropractic Manual treatment + home exercise (procedure+behavior) — The number of treatments will be determined by the individual chiropractor. Chiropractic manual treatment will be limited to gentle spinal manipulation, mobilization and flexion-distraction therapy with light soft tissue massage as indicated to facilitate the manual therapy.
  Patients will attend 4, 45-minute small-group sessions at weeks 1, 2, 4 and 8. At the first two sessions they will be given information about low back pain and shown exercises to perform at home. Emphasis will be placed on the importance of staying active.
  Arms: 1
Procedure: Supervised rehabilitative exercise+home exercise — The rehabilitative exercise program will consist of 20, 1-hour sessions. It is a modification of exercise protocols used in previous studies by the investigators and incorporates recommendations of leading rehabilitative exercise specialists.
  Patients will attend 4, 45-minute small-group sessions at weeks 1, 2, 4 and 8. At the first two sessions they will be given information about low back pain and shown exercises to perform at home. Emphasis will be placed on the importance of staying active.
  Arms: 2
Behavioral: Home exercise — Patients will attend 4, 45-minute small-group sessions at weeks 1, 2, 4 and 8. At the first two sessions they will be given information about low back pain and shown exercises to perform at home. Emphasis will be placed on the importance of staying active.
  Arms: 3

SUMMARY:
The purpose of this randomized clincal trial is to assess the relative effectiveness of three conservative treatment approaches for seniors with chronic low back pain: 1) chiropractic manual treatment plus home exercise, 2) supervised exercise plus home exercise and 3) home exercise alone.

DETAILED DESCRIPTION:
Low back pain (LBP) is a significant health problem for both young and geriatric individuals. Of particular concern is that conditions associated with LBP, such as impaired strength and flexibility, can have very serious consequences for an older individual's independence and overall health.

The broad, long-term objective of this research is to identify effective therapies for low back pain (LBP) and to discover the best methods for enhancing health and functional capacity in the elderly population. This study is a multi-methods clinical trial consisting of a randomized clinical trial (RCT), a cost-effectiveness study alongside the RCT, and a qualitative study nested in the RCT.

This trial builds upon a previous study of chiropractic and exercise funded by HRSA, and focuses on elderly patients with sub-acute and chronic low back pain.

PRIMARY AIMS

* To determine the relative clinical effectiveness the following treatments for LBP patients 65 years and older in both the short-term (after 12 weeks) and long-term (after 52 weeks), using low back pain as the main outcome measure

  1. chiropractic manual treatment plus home exercise
  2. supervised rehabilitative exercise plus home exercise
  3. home exercise

     SECONDARY AIMS
* To estimate the short- and long-term relative effectiveness of the three interventions using:
* Patient-rated outcomes: low back disability, general health status, patient satisfaction, improvement, and medication use measured by self-report questionnaires
* Objective functional performance outcomes: spinal motion, trunk strength and endurance, and functional ability measured by examiners masked to treatment group assignment
* Cost measures: direct and indirect costs of treatment measured by questionnaires, phone interviews, and medical records.
* To describe elderly LBP patients' perceptions of treatment and the issues they consider when determining their satisfaction with care using qualitative methods nested within the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Sub-Acute and chronic low back pain (Defined as current episode more than 6 weeks duration.)
* Quebec Task Force classifications 1, 2, 3 and 4. (This includes patients with back pain, stiffness or tenderness, with or without musculoskeletal signs and neurological signs.{1570})
* 65 years of age and older
* Independent ambulation
* Community dwelling (residency outside nursing home)
* Score of 20 or more on Folstein Mini-Mental State Examination{13246}
* Stable prescription medication plan (no changes in prescription medications that affect musculoskeletal pain in previous month)

Exclusion Criteria:

* Referred low back pain from local joint lesions of the lower extremities or from visceral diseases
* Significant infectious disease Determined by history or by referral to supplementary diagnostic tests
* Ongoing treatment for low back pain by other health care providers
* Mean baseline low back pain score of 20 percentage points or less
* Contraindications to exercise Determined by history or by referral to supplementary diagnostic tests (i.e., uncontrolled arrhythmias, third degree heart block, recent ECG changes, unstable angina, acute myocardial infarction, acute congestive heart failure, cardiomyopathy, valvular heart disease, poorly controlled blood pressure, uncontrolled metabolic disease
* Contraindications to spinal manipulation (i.e. Progressive neurological deficits blood clotting disorders; infectious and non-infectious inflammatory or destructive tissue changes of the spine; severe osteoporosis)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2003-10; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Patient-rated pain (0-11 box scale) | short term = 12 weeks; long term = 52 weeks

SECONDARY OUTCOMES:
General Health | short term = 12 weeks; long term = 52 weeks
Disability | short term = 12 weeks; long term = 52 weeks
Improvement | short term = 12 weeks; long term = 52 weeks
Satisfaction | short term = 12 weeks; long term = 52 weeks
Medication use | short term = 12 weeks; long term = 52 weeks
Biomechanical test: Lumbar spinal motion Trunk strength & endurance Functional Ability Observed Pain Behavior | short term = 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, PhD, Principal Investigator — Northwestern Health Sciences University; Roni Evans, MS, Study Director — Northwestern Health Sciences University
Locations (1):
- Wolfe-Harris Center for Clinical Studies, Northwestern Health Sciences University, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Schulz C, Evans R, Maiers M, Schulz K, Leininger B, Bronfort G. Spinal manipulative therapy and exercise for older adults with chronic low back pain: a randomized clinical trial. Chiropr Man Therap. 2019 May 15;27:21. doi: 10.1186/s12998-019-0243-1. eCollection 2019. PMID 31114673
- [Derived] Maiers MJ, Hartvigsen J, Schulz C, Schulz K, Evans RL, Bronfort G. Chiropractic and exercise for seniors with low back pain or neck pain: the design of two randomized clinical trials. BMC Musculoskelet Disord. 2007 Sep 18;8:94. doi: 10.1186/1471-2474-8-94. PMID 17877825
- See also: Click here for a description of the Wolfe-Harris for Center for Clinical Studies — http://www.nwhealth.edu/research/WHCCS/